CLINICAL TRIAL: NCT01370967
Title: Gastrointestinal Tolerance And General Health Status Of Healthy Term Infants Fed A New Infant Formula: A Prospective, Observational Cohort Study In China
Brief Title: Gastrointestinal Tolerance And General Health Status Of Healthy Term Infants Fed A New Infant Formula
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: B3611002
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: infant; term birth; human milk; infant formula; breast feeding; bottle feeding; gastrointestinal tract; quality of life; infant development
MeSH Terms: conditions — Breast Feeding; Bottle Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Study formula-fed only
  Interventions: Other: Study formula feeding
- Human milk-fed only
  Interventions: Other: Human milk feeding
- Mixed-fed using study formula only
  Interventions: Other: Mixed feeding

INTERVENTIONS:
Other: Study formula feeding — Infants who are exclusively fed the new study formula at time of enrollment
  Groups: Study formula-fed only
Other: Human milk feeding — Infants who are exclusively fed human milk at time of enrollment
  Groups: Human milk-fed only
Other: Mixed feeding — Infants who are exclusively fed human milk and the new study formula at time of enrollment
  Groups: Mixed-fed using study formula only

SUMMARY:
The purpose of this study is to assess stool consistency, in combination with additional health-related parameters including gastrointestinal tolerance and health-related quality of life, in a large sample of Chinese infants. We will also assess the timing of, frequency, and reasons for changes in the choice of formula or method of feeding among infants in this sample, as well as incidence of common infant illness and associated healthcare usage. Anthropometric measures and the frequency and duration of physician- and parent-reported gastrointestinal and other adverse events will be evaluated.

DETAILED DESCRIPTION:
Parents / legally acceptable representatives of eligible infants will be invited to volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term (37-42 weeks gestation), singleton infant at birth.
* Post-natal age between 35 and 49 days (date of birth = day 0) at time of study entry.
* At enrollment, weight-for-age ≥ 5th and ≤ 95th percentile according to World Health Organization growth tables / charts.

Exclusion Criteria:

* Infants who are consuming any types/brands of formula other than the new study formula (either exclusively or in a mixed feeding regimen) at time of study enrollment.
* Suspected or documented severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results, and in the judgment of the investigator, would make the infant inappropriate for entry into the study.

Ages: 35 Days to 49 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy term infants aged approximately 42 days (range 35 - 49 days) who are brought to the health clinic for their first normally-scheduled well-baby visit (i.e. typically age 42 days in China).
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Infant stool consistency and frequency (assessed using a 3-day stool diary) | Baseline
Infant stool consistency and frequency (assessed using a 3-day stool diary) | day 15
Infant stool consistency and frequency (assessed using a 3-day stool diary) | day 30
Infant stool consistency and frequency (assessed using a 3-day stool diary) | day 45

SECONDARY OUTCOMES:
Infant gastrointestinal tolerance (assessed using a validated, interviewer-assisted parent questionnaire) | Baseline
Infant gastrointestinal tolerance (assessed using a validated, interviewer-assisted parent questionnaire) | day 18
Infant gastrointestinal tolerance (assessed using a validated, interviewer-assisted parent questionnaire) | day 48
Infant and parent health-related quality of life (assessed using validated parent questionnaires) | Baseline
Infant and parent health-related quality of life (assessed using validated parent questionnaires) | day 48

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - The 306th Hospital of PLA, Chaoyang District, Beijing Municipality
  - Beijing Haidian Maternal&Child Health Hospital, Haidian District, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Yuzhong, Chongqing Municipality
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhu Jiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Zhongshan Bo'ai Hospital, Zhongshan, Guangdong
  - Changsha Hospital for Maternal&Child Health Care, Changsha, Hunan
  - Maternity and Child Health Care Hospital in Jiangsu Province, Nanjing, Jiangsu
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Chengdu Women & Children Center Hospital, Chengdu, Sichuan
  - West China Second University Hospital, SCU, Chengdu, Sichuan
  - Tianjin First Center Hospital, Nankai, Tianjin Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Ningbo Yinzhou People's Hospital, Ningbo, Zhejiang
  - Beijing Obstetrics Gynecology Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Shanghai Children's Medical Center Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Children's Hospital of Fudan University, Shanghai

REFERENCES:
- [Derived] Hays NP, Mao M, Zhang L, Ge J, Northington R, Yao M, Volger S. Infant feeding and health-related quality of life in healthy Chinese infants: results from a prospective, observational cohort study. Health Qual Life Outcomes. 2016 Aug 8;14(1):116. doi: 10.1186/s12955-016-0518-3. PMID 27502768
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3611002&StudyName=Gastrointestinal%20Tolerance%20And%20General%20Health%20Status%20Of%20Healthy%20Term%20Infants%20Fed%20A%20New%20Infant%20Formula